CLINICAL TRIAL: NCT01558505
Title: Drug Eluting Balloon in peripherAl inTErvention For Below The Knee Angioplasty Evaluation: the DEBATE-BTK Study
Brief Title: Drug Eluting Balloon in peripherAl inTErvention For Below The Knee Angioplasty Evaluation
Acronym: DEBATE-BTK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leonardo Bolognese, MD (Other)
Responsible Party: Sponsor-Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Organization: Ospedale San Donato (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arezzo005
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Critical Limb Ischemia
Keywords: critical limb ischemia; drug-eluting balloon; restenosis
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard PTA (Active Comparator): conventional balloon angioplasty
  Interventions: Device: POBA
- Drug-eluting balloon angioplasty (Experimental): paclitaxel-eluting balloon angioplasty
  Interventions: Device: PEB

INTERVENTIONS:
Device: PEB — paclitaxel-eluting balloon angioplasty
  Arms: Drug-eluting balloon angioplasty
Device: POBA — conventional balloon angioplasty
  Arms: standard PTA

SUMMARY:
Drug-eluting balloon showed positive results in terms of restenosis reduction in peripheral intervention (PTA). The aim of the study is to investigate in a randomized fashion the efficacy and safety of Paclitaxel-eluting balloon (PEB) (In.Pact Amphirion, Invatec, Brescia, Italy) versus non drug-eluting balloon (NEB) (Amphirion deep, Invatec, Brescia, Italy) in diabetic patients with Critical Limb Ischemia (CLI) undergoing PTA of below-the-knee (BTK) vessels.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* angiographic stenosis>50% or occlusion of one below-knee vessel

Exclusion Criteria:

* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent
* need for amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
angiographic binary restenosis | 12 months
  incidence of binary restenosis

SECONDARY OUTCOMES:
major amputation | 24 motnhs
  incidence of major amputation
target lesion revascularization | 24 months
  incidence of target lesion revascularization
vessel reocclusion | 24 months
  incidence of vessel reocclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Liistro F, Porto I, Angioli P, Grotti S, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for below the knee angioplasty evaluation (DEBATE-BTK): a randomized trial in diabetic patients with critical limb ischemia. Circulation. 2013 Aug 6;128(6):615-21. doi: 10.1161/CIRCULATIONAHA.113.001811. PMID 23797811